CLINICAL TRIAL: NCT05614960
Title: The Bioavailability of Vitamin B12 From Nori in Vegetarians: a Dose Response Study
Brief Title: Dried Purple Laver (Nori) as a Food Source of Vitamin B12 in Vegetarians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Tina Hsueh-Ting Chiu, Associate Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FuJenCU
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Vitamin B12; Vegetarian diet; Purple laver (Porphyra sp.); Nori
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2.4μg vitamin B12 (Experimental): Participants need to consume 4 sheets (5g) of dried purple laver (Nori) daily for 4 weeks.
  Interventions: Other: Dried purple laver (Nori)
- 4μg vitamin B12 (Experimental): Participants need to consume 7 sheets (8g) of dried purple laver (Nori) daily for 4 weeks.
  Interventions: Other: Dried purple laver (Nori)
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Dried purple laver (Nori) — Dried purple laver (Nori) that has been test to have bioactivity vitamin B12 will be given for intervention groups.
  Arms: 2.4μg vitamin B12; 4μg vitamin B12

SUMMARY:
This is an intervention study aiming to understand the bioavailability of vitamin B12 from nori for vegetarians.

DETAILED DESCRIPTION:
Thirty vegetarian participants will be randomly assigned to one of three intervention arms: (1) 5g of nori (4 sheets, containing 2.4μg vitamin B12), (2) 8g nori (7 sheets, containing 4μg vitamin B12), (3) control group (no nori). At baseline and end of 4 weeks, participants will be measured on serum vitamin B12, methylmalonic acid, holotranscobalamin, homocysteine and folate.

ELIGIBILITY:
Inclusion Criteria:

* Vegetarians (including vegan, ovo-vegetarian, lacto-vegetarian, lacto-ovo vegetarian)
* Duration of the vegetarian diet: at least 1 year
* Aged 20-60 years old
* Have not taken vitamin B12 or folate supplement within 1 year
* Willing to adhere to study intervention and be tested for vitamin B12 related biomarkers.
* Familiar with LINE application on smartphone

Exclusion Criteria:

* Any disease or surgery that affects the vitamin B12 status (Pernicious anemia, Gastrointestinal disease and surgery, Pancreatic diseases, Chronic kidney disease)
* Hyperthyroidism
* Previous adverse reaction to nori
* Have taken antacid or metformin in the past 1 week
* Alcoholic and not willing to abstinence from alcoholic beverages

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in holotranscobalamin in 4 weeks | 4 weeks (Week 4 - Baseline)
  Assessing the change in serum holotranscobalamin after consuming varying doses of nori
Change in methylmalonic acid in 4 weeks | 4 weeks (Week 4 - Baseline)
  Assessing the change in serum methylmalonic acid after consuming varying doses of nori

SECONDARY OUTCOMES:
Change in serum vitamin B12 concentration in 4 weeks | 4 weeks (Week 4 - Baseline)
  Assessing the change in serum vitamin B12 after consuming varying doses of nori
Change in homocysteine in 4 weeks | 4 weeks (Week 4 - Baseline)
  Assessing the change in serum homocysteine after consuming varying doses of nori

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hsueh-Ting Chiu, PhD, Principal Investigator — Fu-Jen Catholic University, Department of Nutritional Science
Locations (1):
- Department of Nutritional Science, Fu-Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu THT, Kao YC, Wang LY, Chang HR, Lin CL. A Dietitian-Led Vegan Program May Improve GlycA, and Other Novel and Traditional Cardiometabolic Risk Factors in Patients With Dyslipidemia: A Pilot Study. Front Nutr. 2022 Mar 24;9:807810. doi: 10.3389/fnut.2022.807810. eCollection 2022. PMID 35399690
- [Background] Takenaka S, Sugiyama S, Ebara S, Miyamoto E, Abe K, Tamura Y, Watanabe F, Tsuyama S, Nakano Y. Feeding dried purple laver (nori) to vitamin B12-deficient rats significantly improves vitamin B12 status. Br J Nutr. 2001 Jun;85(6):699-703. doi: 10.1079/bjn2001352. PMID 11430774
- [Background] Suzuki H. Serum vitamin B12 levels in young vegans who eat brown rice. J Nutr Sci Vitaminol (Tokyo). 1995 Dec;41(6):587-94. doi: 10.3177/jnsv.41.587. PMID 8926531
- [Background] Schwarz J, Dschietzig T, Schwarz J, Dura A, Nelle E, Watanabe F, Wintgens KF, Reich M, Armbruster FP. The influence of a whole food vegan diet with Nori algae and wild mushrooms on selected blood parameters. Clin Lab. 2014;60(12):2039-50. doi: 10.7754/clin.lab.2014.140527. PMID 25651739
- [Background] Rauma AL, Torronen R, Hanninen O, Mykkanen H. Vitamin B-12 status of long-term adherents of a strict uncooked vegan diet ("living food diet") is compromised. J Nutr. 1995 Oct;125(10):2511-5. doi: 10.1093/jn/125.10.2511. PMID 7562085
- [Background] Watanabe F, Yabuta Y, Bito T, Teng F. Vitamin B(1)(2)-containing plant food sources for vegetarians. Nutrients. 2014 May 5;6(5):1861-73. doi: 10.3390/nu6051861. PMID 24803097
- [Background] Rizzo G, Lagana AS, Rapisarda AM, La Ferrera GM, Buscema M, Rossetti P, Nigro A, Muscia V, Valenti G, Sapia F, Sarpietro G, Zigarelli M, Vitale SG. Vitamin B12 among Vegetarians: Status, Assessment and Supplementation. Nutrients. 2016 Nov 29;8(12):767. doi: 10.3390/nu8120767. PMID 27916823
- [Derived] Huang QN, Watanabe F, Koseki K, He RE, Lee HL, Chiu THT. Effect of roasted purple laver (nori) on vitamin B12 nutritional status of vegetarians: a dose-response trial. Eur J Nutr. 2024 Dec;63(8):3269-3279. doi: 10.1007/s00394-024-03505-9. Epub 2024 Oct 1. PMID 39352476